CLINICAL TRIAL: NCT00568945
Title: Study to Investigate the Effect of the A1 Agonist Capadenoson on Ventricular HR in Patients With Persistent or Permanent Atrial Fibrillation by Administration of Capadenoson in a Dose of 4 mg Once Daily for Five Days
Brief Title: Study to Investigate the Effect of the A1 Agonist Capadenoson on Ventricular HR in Patients With Persistent or Permanent Atrial Fibrillation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12679; 2007-003619-30 (EudraCT Number)
Record Dates: First submitted 2007-10-25; First posted 2007-12-06 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Capadenoson
MeSH Terms: conditions — Atrial Fibrillation | interventions — capadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Capadenoson (BAY68-4986)

INTERVENTIONS:
Drug: Capadenoson (BAY68-4986) — 4 mg BAY68-4986 for five days

SUMMARY:
This trial has the primary goal to show that BAY68-4986 can lower the ventricular rate in patients with the indication persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female (without childbearing potential) white patients
* History of persistent or permanent atrial fibrillation
* 18 to 75 years of age

Exclusion Criteria:

* Patients with high-risk cardiovascular diseases
* Stroke or myocardial infarction
* Relevant pathological changes in the ECG or echocardiography
* Medication affecting ventricular response in Afib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The effect of capadenoson (BAY68-4986) on rate control in patients with atrial fibrillation | 1 week

SECONDARY OUTCOMES:
To investigate safety and tolerability of this treatment with capadenoson | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Erfurt, Thuringia, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/